CLINICAL TRIAL: NCT01874431
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Safety and Efficacy of Different Oral Doses of BAY94-8862 in Subjects With Type 2 Diabetes Mellitus and the Clinical Diagnosis of Diabetic Nephropathy
Brief Title: Safety and Efficacy of Different Oral Doses of BAY94-8862 in Subjects With Type 2 Diabetes Mellitus and the Clinical Diagnosis of Diabetic Nephropathy
Acronym: ARTS-DN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16243; 2012-004179-38 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Finerenone (BAY94-8862) (1.25 mg) (Experimental): 1.25 mg dose oral once daily for 90 days
  Interventions: Drug: Finerenone (BAY94-8862)
- Finerenone (BAY94-8862)(2.5 mg) (Experimental): 2.5 mg dose oral once daily for 90 days
  Interventions: Drug: Finerenone (BAY94-8862)
- Finerenone (BAY94-8862)(5 mg) (Experimental): 5 mg dose oral once daily for 90 days
  Interventions: Drug: Finerenone (BAY94-8862)
- Finerenone (BAY94-8862)(7.5 mg) (Experimental): 7.5 mg dose oral once daily for 90 days
  Interventions: Drug: Finerenone (BAY94-8862)
- Finerenone (BAY94-8862) (10 mg) (Experimental): 10 mg dose oral once daily for 90 days
  Interventions: Drug: Finerenone (BAY94-8862)
- Finerenone (BAY94-8862) (15 mg) (Experimental): 15 mg dose oral once daily for 90 days
  Interventions: Drug: Finerenone (BAY94-8862)
- Finerenone (BAY94-8862)(20 mg) (Experimental): 20 mg dose oral once daily for 90 days
  Interventions: Drug: Finerenone (BAY94-8862)
- Placebo (Placebo Comparator): Placebo oral dose once daily for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY94-8862)
  Arms: Finerenone (BAY94-8862) (1.25 mg); Finerenone (BAY94-8862) (10 mg); Finerenone (BAY94-8862) (15 mg); Finerenone (BAY94-8862)(2.5 mg); Finerenone (BAY94-8862)(20 mg); Finerenone (BAY94-8862)(5 mg); Finerenone (BAY94-8862)(7.5 mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess a new drug, BAY94-8862 given orally at different doses, to evaluate whether it was safe and can help the well being of patients with type 2 diabetes and diabetic nephropathy. These treatment doses were compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older.The lower age limit may be higher if legally required in the participating country
* Women of childbearing potential can only be included in the study if a pregnancy test is negative and if they agree to use adequate contraception when sexually active.
* Subjects with type 2 diabetes mellitus fulfilling at least 1 of the following criteria

  * are on oral antidiabetics and / or insulin,
  * have a documented fasting glucose >/= 7.0 mmol/L in the medical history,
  * have a 2 hour plasma glucose >/=11.1 mmol/L during an oral glucose tolerance test in the medical history, or
  * have a glycated hemoglobin (HbA1c) >/=6.5% [National Glycohemoglobin Standardization Program (NGSP) / Diabetes Control and Complications Trial (DCCT)] in the medical history or at the run-in visit
* Subjects with a clinical diagnosis of diabetic nephropathy (DN) based on at least 1 of the following criteria:

  * Persistent very high albuminuria defined as urinary albumin-to-creatine ratio (UACR) of >/=300 mg/g ( >/= 34 mg/mmol) in 2 out of 3 first morning void samples and estimated glomerular filtration rate (eGFR) >/=30 mL/min/1.73 m² but < 90 mL/min/1.73m² (Chronic Kidney Disease Epidemiology Collaboration, CKD EPI) (mL = milliliter; min = minute; m2 = square meter; g = gram; mmol = millimole) or
  * Persistent high albuminuria defined as UACR of >/=30 mg/g but <300 mg/g in (>/=3.4mg/mmol but <34 mg/mmol) in 2 out of 3 first morning void samples and eGFR >/=30 mL/min/1.73 m² but < 90 mL/min/1.73m²
* Subjects treated with an angiotensin-converting enzyme inhibitor (ACEI) and/or angiotensin receptor blocker (ARB) for at least 3 months without any adjustments to this therapy for at least 4 weeks prior to the screening visit
* Serum potassium </= 4.8 mmol/L at both the run-in visit and the screening visit

Exclusion Criteria:

* Non-diabetic renal disease
* Glycated hemoglobin (HbA1c) >12% at the run-in visit or the screening visit
* UACR >3000 mg/g (339mg/mmol) in any of the urinary first morning void samples at the run-in visit or screening visit
* Hypertension with mean sitting systolic blood pressure (SBP) >/=180 mmHg or mean sitting diastolic blood pressure (DBP) >/=110 mmHg at the run-in visit or mean supine SBP >/=160 mmHg or mean sitting DBP >/=100 mmHg at the screening visit
* Subjects with a clinical diagnosis of heart failure with reduced ejection fraction (HFrEF) and persistent symptoms (New York Heart Association class II-IV) at the run-in visit
* Concomitant therapy with eplerenone, spironolactone, any renin inhibitor, or potassium-sparing diuretic
* Dialysis for acute renal failure within the previous 6 months prior to the run-in visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2014-07-09 (Actual); Study Completion 2014-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (130):
- United States (14):
  - Birmingham, Alabama
  - Chula Vista, California
  - Los Angeles, California
  - Los Gatos, California
  - New Haven, Connecticut
  - Miami, Florida
  - Pembroke Pines, Florida
  - Chicago, Illinois
  - Flint, Michigan
  - Flushing, New York
  - Orangeburg, South Carolina
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Burlington, Vermont
- Australia (7):
  - St Leonards, New South Wales
  - Clayton, Victoria
  - Melbourne, Victoria
  - Prahran, Victoria
  - Reservoir, Victoria
  - Box Hill
  - Woolloongabba
- Austria (5):
  - Graz
  - Innsbruck
  - Salzburg
  - Sankt Pölten
  - Vienna
- Bulgaria (7):
  - Haskovo
  - Lukovit
  - Plovdiv
  - Rousse
  - Sofia
  - Stara Zagora
  - Varna
- Canada (6):
  - Vancouver, British Columbia
  - Courtice, Ontario
  - Kitchener, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (4):
  - Chrudim
  - Kopřivnice
  - Krnov
  - Prague
- Denmark (7):
  - Aarhus C
  - Gentofte Municipality
  - Herlev
  - Hillerød
  - Holbæk
  - Holstebro
  - Kolding
- Finland (5):
  - Helsinki
  - Jyväskylä
  - Oulu
  - Tampere
  - Turku
- France (5):
  - Amiens
  - La Tronche
  - Lyon
  - Paris
  - Strasbourg
- Germany (5):
  - Hanover, Lower Saxony
  - Bad Oeynhausen, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Neuwied, Rhineland-Palatinate
- Hong Kong (2):
  - Hong Kong
  - Shatin
- Hungary (5):
  - Budapest
  - Debrecen
  - Eger
  - Nagykanizsa
  - Pápa
- Israel (6):
  - Ashkelon
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Tel Aviv
- Italy (8):
  - Foggia, Apulia
  - Napoli, Campania
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Monza-Brianza, Lombardy
  - Cagliari, Sardinia
  - Pisa, Tuscany
  - Padua, Veneto
- Netherlands (5):
  - Almere Stad
  - Eindhoven
  - Groningen
  - Hoogeveen
  - Maastricht
- Norway (2):
  - Ålesund
  - Hamar
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Lodz
  - Lublin
  - Oława
  - Warsaw
  - Wroclaw
- Portugal (2):
  - Almada
  - Lisbon
- South Africa (11):
  - Klipsruit West, Gauteng
  - Krugersdorp, Gauteng
  - Lenasia South, Gauteng
  - Newtown, Gauteng
  - Durban, KwaZulu-Natal
  - Merebank, KwaZulu-Natal
  - Tongaat, KwaZulu-Natal
  - Cape Town, Western Cape
  - Goodwood, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
- South Korea (2):
  - Busan
  - Seoul
- Spain (6):
  - Ferrol, A Coruña
  - Jerez de la Frontera, Cádiz
  - Sagunto, Valencia
  - Barcelona
  - Girona
  - Madrid
- Sweden (7):
  - Karlstad
  - Kristianstad
  - Örebro
  - Skövde
  - Stockholm
  - Uppsala
  - Vällingby
- Taiwan (2):
  - Kaohsiung City
  - Taipei

REFERENCES:
- [Result] Bakris GL, Agarwal R, Chan JC, Cooper ME, Gansevoort RT, Haller H, Remuzzi G, Rossing P, Schmieder RE, Nowack C, Kolkhof P, Joseph A, Pieper A, Kimmeskamp-Kirschbaum N, Ruilope LM; Mineralocorticoid Receptor Antagonist Tolerability Study-Diabetic Nephropathy (ARTS-DN) Study Group. Effect of Finerenone on Albuminuria in Patients With Diabetic Nephropathy: A Randomized Clinical Trial. JAMA. 2015 Sep 1;314(9):884-94. doi: 10.1001/jama.2015.10081. PMID 26325557
- [Result] Snelder N, Heinig R, Drenth HJ, Joseph A, Kolkhof P, Lippert J, Garmann D, Ploeger B, Eissing T. Population Pharmacokinetic and Exposure-Response Analysis of Finerenone: Insights Based on Phase IIb Data and Simulations to Support Dose Selection for Pivotal Trials in Type 2 Diabetes with Chronic Kidney Disease. Clin Pharmacokinet. 2020 Mar;59(3):359-370. doi: 10.1007/s40262-019-00820-x. PMID 31583611
- [Result] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Ostrominski JW, Filippatos G, Claggett BL, Miao ZM, Desai AS, Jhund PS, Henderson A, Rohwedder K, Brinker MD, Scalise A, Schloemer P, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Rossing P, Ruilope LM, Anker SD, Pitt B, Agarwal R, McMurray JJV, Solomon SD, Vaduganathan M. Effect of Finerenone on Morbidity and Mortality in CKD. J Am Soc Nephrol. 2025 Sep 12. doi: 10.1681/ASN.0000000823. Online ahead of print. No abstract available. PMID 40938666
- [Derived] Agarwal R, Ruilope LM, Ruiz-Hurtado G, Haller H, Schmieder RE, Anker SD, Filippatos G, Pitt B, Rossing P, Lambelet M, Nowack C, Kolkhof P, Joseph A, Bakris GL. Effect of finerenone on ambulatory blood pressure in chronic kidney disease in type 2 diabetes. J Hypertens. 2023 Feb 1;41(2):295-302. doi: 10.1097/HJH.0000000000003330. Epub 2022 Dec 8. PMID 36583355
- [Derived] Erraez S, Lopez-Mesa M, Gomez-Fernandez P. Mineralcorticoid receptor blockers in chronic kidney disease. Nefrologia (Engl Ed). 2021 May-Jun;41(3):258-275. doi: 10.1016/j.nefro.2020.10.001. Epub 2020 Dec 24. English, Spanish. PMID 33358451
- See also: Click here to find results for studies related to Bayer Healthcare products. — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 148 study centers in 23 countries, from 12 June 2013 (first participant, first visit) to 07 August 2014 (last participant, last visit). The randomization was stratified by region (Europe, North America, Asia, others [Australia, Israel, and South Africa]), and type of albuminuria at screening (very high or high albuminuria).
Pre-assignment Details: Of 1501 participants screened, 823 were randomized at 128 study centers and 678 were screening failures. The reasons were not fulfilled inclusion-/exclusion criteria's (635 participants), withdrawal by participants (37 participants), adverse event (3 participants), physician decision (2 participants), logistical difficulties (1 participant) and lost to follow-up (1 participant).
Groups:
- Finerenone (BAY94-8862) (1.25 mg): 1.25 milligram (mg) BAY94-8862 tablet once daily in the morning for 90 days.
- Finerenone (BAY94-8862) (2.5 mg): 2.5 mg BAY94-8862 tablet once daily in the morning for 90 days.
- Finerenone (BAY94-8862) (5 mg): 5 mg BAY94-8862 tablet once daily in the morning for 90 days.
- Finerenone (BAY94-8862) (7.5 mg): 7.5 mg BAY94-8862 tablet once daily in the morning for 90 days.
- Finerenone (BAY94-8862) (10 mg): 10 mg BAY94-8862 tablet once daily in the morning for 90 days.
- Finerenone (BAY94-8862) (15 mg): 15 mg BAY94-8862 tablet once daily in the morning for 90 days.
- Finerenone (BAY94-8862) (20 mg): 20 mg BAY94-8862 tablet once daily in the morning for 90 days
- Placebo: Placebo tablet once daily in the morning for 90 days.
Period: Overall Study
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862) (2.5 mg) | Finerenone (BAY94-8862) (5 mg) | Finerenone (BAY94-8862) (7.5 mg) | Finerenone (BAY94-8862) (10 mg) | Finerenone (BAY94-8862) (15 mg) | Finerenone (BAY94-8862) (20 mg) | Placebo
Started | 96 | 92 | 100 | 98 | 98 | 125 | 120 | 94
Participants Received Treatment | 96 | 92 | 100 | 97 | 98 | 125 | 119 | 94
Completed | 90 | 87 | 90 | 91 | 90 | 114 | 112 | 90
Not Completed | 6 | 5 | 10 | 7 | 8 | 11 | 8 | 4
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 6 | 5 | 2 | 8 | 2 | 3
Not completed — Protocol Violation | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 1
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Logistical difficulties | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 0
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): all randomized subjects who took at least one dose of study drug and with data after beginning of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862) (2.5 mg) | Finerenone (BAY94-8862) (5 mg) | Finerenone (BAY94-8862) (7.5 mg) | Finerenone (BAY94-8862) (10 mg) | Finerenone (BAY94-8862) (15 mg) | Finerenone (BAY94-8862) (20 mg) | Placebo | Total
Number analyzed (Participants) | 96 | 92 | 100 | 97 | 98 | 125 | 119 | 94 | 821
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.91 (9.57) | 64.86 (9.09) | 63.31 (8.79) | 63.73 (10.04) | 64.94 (9.62) | 63.95 (8.34) | 64.70 (9.26) | 63.26 (8.68) | 64.21 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 29 | 18 | 21 | 27 | 30 | 25 | 182
  Male | 78 | 78 | 71 | 79 | 77 | 98 | 89 | 69 | 639
Baseline UACR [Mean (Standard Deviation); unit: g/kg] — Albumin-to-creatinine ratio (UACR) is defined as gram of albumin per kilogram of creatinine. UACR was determined from 3 first morning void samples taken on 3 consecutive days.
  g/kg | 412.02 (507.51) | 471.01 (784.84) | 402.04 (535.44) | 405.14 (702.63) | 441.16 (571.27) | 450.12 (657.04) | 379.28 (457.33) | 377.28 (542.27) | 417.16 (599.12)
Baseline potassium [Mean (Standard Deviation); unit: mmol/L] | 4.323 (0.425) | 4.297 (0.426) | 4.314 (0.325) | 4.311 (0.435) | 4.297 (0.420) | 4.288 (0.459) | 4.294 (0.439) | 4.254 (0.479) | 4.297 (0.427)
Baseline eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] — An estimated glomerular filtration rate (eGFR) indicates the renal function. An eGFR was calculated based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
  mL/min/1.73m^2 | 66.113 (21.923) | 67.425 (20.164) | 67.080 (22.205) | 67.497 (21.917) | 67.042 (20.857) | 67.455 (23.646) | 66.039 (22.205) | 72.213 (20.434) | 67.544 (21.772)
Baseline KDQOL-36 domain score (Effects of Kidney Disease) [Mean (Standard Deviation); unit: Scores on a scale] — The Kidney Disease QOL [KDQOL]-36 questionnaire is a specific measure of Health-Related Quality of Life (HRQoL) for chronic kidney disease (CKD) that includes effects and burden of kidney disease as well as physical and mental health scores. Index score ranges from 0 (serve problems in all items) to 100 (no problem in all items). "Effects of Kidney disease" subscore was analyzed. Population: Participants with valid data for this baseline characteristic
  Scores on a scale
    number analyzed (Participants) | 95 | 90 | 97 | 96 | 96 | 122 | 116 | 93 | 805
    (all) | 90.78 (10.28) | 92.53 (9.57) | 91.78 (12.55) | 92.99 (11.04) | 88.71 (16.50) | 90.45 (14.39) | 89.10 (17.45) | 81.45 (20.42) | 90.57 (13.69)
Baseline EQ-5D scores (EQ5D - Visual Analog Scale) [Mean (Standard Deviation); unit: Score on a scale] — EuroQol Group 5-Dimension, 3-Level (EQ-5D-3L) questionnaires consist of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS was analyzed for this endpoint and it ranges from 0 (worst possible health state) to 100 (best possible health state). Population: Participants with valid data for this baseline characteristic
  Score on a scale
    number analyzed (Participants) | 96 | 89 | 95 | 96 | 95 | 121 | 117 | 92 | 801
    (all) | 71.76 (16.39) | 72.79 (14.81) | 73.01 (16.21) | 74.49 (15.92) | 73.89 (16.47) | 73.19 (16.11) | 71.36 (17.49) | 70.05 (17.69) | 72.56 (16.42)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of UACR at Day 90 to UACR at Baseline
Description: Albumin-to-creatinine ratio (UACR) is defined as gram of albumin per kilogram of creatinine. UACR was calculating the average of 3 first morning void samples taken on 3 consecutive days.
Time Frame: Baseline and Day 90±2
Population: Full analysis set (FAS): included all participants of the SAF who had baseline and at least one post-baseline UACR value.
Measure: Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862) (2.5 mg) | Finerenone (BAY94-8862) (5 mg) | Finerenone (BAY94-8862) (7.5 mg) | Finerenone (BAY94-8862) (10 mg) | Finerenone (BAY94-8862) (15 mg) | Finerenone (BAY94-8862) (20 mg) | Placebo
Number analyzed (Participants) | 96 | 92 | 98 | 96 | 96 | 123 | 117 | 94
Ratio | 0.869 (0.772) [0.772 to 0.979] | 0.89 (0.786) [0.786 to 1.009] | 0.824 (0.73) [0.73 to 0.929] | 0.739 (0.653) [0.653 to 0.835] | 0.708 (0.627) [0.627 to 0.8] | 0.63 (0.563) [0.563 to 0.705] | 0.585 (0.523) [0.523 to 0.654] | 0.938 (0.829) [0.829 to 1.061]
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) (1.25 mg) vs Placebo; To demonstrate a dose-dependent effect of finerenone, an analysis of covariance (ANCOVA) with factors treatment group, type of albuminuria at screening and region, and log-transformed baseline value as covariate nested within type of albuminuria at screening was performed in the FAS using a last-observation carried-forward (LOCF) method for missing observations; Test type: Other; p = 0.1973, t-test, 1 sided; Least square mean ratio = 0.926, 90% CI 2-sided [0.799 to 1.074]
Statistical Analysis 2: Comparison: Finerenone (BAY94-8862) (2.5 mg) vs Placebo; To demonstrate a dose-dependent effect of finerenone, an ANCOVA with factors treatment group, type of albuminuria at screening and region, and log-transformed baseline value as covariate nested within type of albuminuria at screening was performed in the FAS using a LOCF method for missing observations; Test type: Other; p = 0.2808, t-test, 1 sided; Least square mean ratio = 0.949, 90% CI 2-sided [0.818 to 1.101]
Statistical Analysis 3: Comparison: Finerenone (BAY94-8862) (5 mg) vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.0723, t-test, 1 sided; Least square mean ratio = 0.878, 90% CI 2-sided [0.758 to 1.017]
Statistical Analysis 4: Comparison: Finerenone (BAY94-8862) (7.5 mg) vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.0039, t-test, 1 sided; Least square mean ratio = 0.787, 90% CI 2-sided [0.68 to 0.912]
Statistical Analysis 5: Comparison: Finerenone (BAY94-8862) (10 mg) vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.0009, t-test, 1 sided; Least square mean ratio = 0.755, 90% CI 2-sided [0.651 to 0.875]
Statistical Analysis 6: Comparison: Finerenone (BAY94-8862) (15 mg) vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p < 0.0001, t-test, 1 sided; Least square mean ratio = 0.671, 90% CI 2-sided [0.584 to 0.772]
Statistical Analysis 7: Comparison: Finerenone (BAY94-8862) (20 mg) vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p < 0.0001, t-test, 1 sided; Least square mean ratio = 0.624, 90% CI 2-sided [0.542 to 0.718]

2. Secondary Outcome: Change From Baseline to Day 90 in Serum Potassium
Time Frame: Baseline and Day 90±2
Population: Participants in SAF with valid data for this endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862) (2.5 mg) | Finerenone (BAY94-8862) (5 mg) | Finerenone (BAY94-8862) (7.5 mg) | Finerenone (BAY94-8862) (10 mg) | Finerenone (BAY94-8862) (15 mg) | Finerenone (BAY94-8862) (20 mg) | Placebo
Number analyzed (Participants) | 90 | 87 | 85 | 88 | 87 | 109 | 112 | 90
millimole per liter | 0.109 [0.030 to 0.187] | 0.123 [0.043 to 0.203] | 0.202 [0.122 to 0.282] | 0.127 [0.047 to 0.207] | 0.167 [0.087 to 0.248] | 0.238 [0.165 to 0.31] | 0.188 [0.116 to 0.259] | 0.002 [-0.077 to 0.081]
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) (1.25 mg) vs Placebo; Test type: Other; p = 0.0428, t-test, 2 sided; Least squares mean difference = 0.107, 95% CI 2-sided [0.003 to 0.21]
Statistical Analysis 2: Comparison: Finerenone (BAY94-8862) (2.5 mg) vs Placebo; Test type: Other; p = 0.0223, t-test, 2 sided; Least squares mean difference = 0.121, 95% CI 2-sided [0.017 to 0.225]
Statistical Analysis 3: Comparison: Finerenone (BAY94-8862) (5 mg) vs Placebo; Test type: Other; p = 0.0002, t-test, 2 sided; Least squares mean difference = 0.2, 95% CI 2-sided [0.096 to 0.305]
Statistical Analysis 4: Comparison: Finerenone (BAY94-8862) (7.5 mg) vs Placebo; Test type: Other; p = 0.0181, t-test, 2 sided; Least squares mean difference = 0.125, 95% CI 2-sided [0.021 to 0.229]
Statistical Analysis 5: Comparison: Finerenone (BAY94-8862) (10 mg) vs Placebo; Test type: Other; p = 0.0019, t-test, 2 sided; Least squares mean difference = 0.166, 95% CI 2-sided [0.061 to 0.27]
Statistical Analysis 6: Comparison: Finerenone (BAY94-8862) (15 mg) vs Placebo; Test type: Other; p < 0.0001, t-test, 2 sided; Least squares mean difference = 0.236, 95% CI 2-sided [0.137 to 0.334]
Statistical Analysis 7: Comparison: Finerenone (BAY94-8862) (20 mg) vs Placebo; Test type: Other; p = 0.0002, t-test, 2 sided; Least squares mean difference = 0.186, 95% CI 2-sided [0.088 to 0.284]

3. Secondary Outcome: Change From Baseline to Day 90 in eGFR
Description: An estimated glomerular filtration rate (eGFR) indicates the renal function. An eGFR was calculated based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
Time Frame: Baseline and Day 90±2
Population: Participants in SAF with valid data for this endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m^2
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862) (2.5 mg) | Finerenone (BAY94-8862) (5 mg) | Finerenone (BAY94-8862) (7.5 mg) | Finerenone (BAY94-8862) (10 mg) | Finerenone (BAY94-8862) (15 mg) | Finerenone (BAY94-8862) (20 mg) | Placebo
Number analyzed (Participants) | 90 | 87 | 85 | 88 | 87 | 113 | 112 | 90
mL/min/1.73m^2 | -2.364 (-4.311) [-4.311 to -0.418] | -3.189 (-5.164) [-5.164 to -1.213] | -2.497 (-4.475) [-4.475 to -0.518] | -3.378 (-5.341) [-5.341 to -1.415] | -4.192 (-6.181) [-6.181 to -2.202] | -3.806 (-5.563) [-5.563 to -2.05] | -4.024 (-5.792) [-5.792 to -2.256] | -1.578 (-3.53) [-3.53 to 0.373]
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) (1.25 mg) vs Placebo; Test type: Other; p = 0.5454, t-test, 2 sided; Least squares mean difference = -0.786, 95% CI 2-sided [-3.337 to 1.765]
Statistical Analysis 2: Comparison: Finerenone (BAY94-8862) (2.5 mg) vs Placebo; Test type: Other; p = 0.2186, t-test, 2 sided; Least squares mean difference = -1.61, 95% CI 2-sided [-4.177 to 0.957]
Statistical Analysis 3: Comparison: Finerenone (BAY94-8862) (5 mg) vs Placebo; Test type: Other; p = 0.4859, t-test, 2 sided; Least squares mean difference = -0.918, 95% CI 2-sided [-3.503 to 1.667]
Statistical Analysis 4: Comparison: Finerenone (BAY94-8862) (7.5 mg) vs Placebo; Test type: Other; p = 0.1677, t-test, 2 sided; Least squares mean difference = -1.8, 95% CI 2-sided [-4.358 to 0.759]
Statistical Analysis 5: Comparison: Finerenone (BAY94-8862) (10 mg) vs Placebo; Test type: Other; p = 0.0462, t-test, 2 sided; Least squares mean difference = -2.613, 95% CI 2-sided [-5.183 to -0.044]
Statistical Analysis 6: Comparison: Finerenone (BAY94-8862) (15 mg) vs Placebo; Test type: Other; p = 0.0705, t-test, 2 sided; Least squares mean difference = -2.228, 95% CI 2-sided [-4.643 to 0.187]
Statistical Analysis 7: Comparison: Finerenone (BAY94-8862) (20 mg) vs Placebo; Test type: Other; p = 0.048, t-test, 2 sided; Least squares mean difference = -2.446, 95% CI 2-sided [-4.869 to -0.022]

4. Secondary Outcome: Change From Baseline to Day 90 in KDQOL-36 Domain Score (Effects of Kidney Disease)
Description: The Kidney Disease QOL [KDQOL]-36 questionnaire is a specific measure of Health-Related Quality of Life (HRQoL) for chronic kidney disease (CKD) that includes effects and burden of kidney disease as well as physical and mental health scores. Index score ranges from 0 (severe problems in all items) to 100 (no problem in all items). "Effects of Kidney disease" subscore was analyzed.
Time Frame: Baseline and Day 90±2
Population: Participants in FAS with valid data for this endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862) (2.5 mg) | Finerenone (BAY94-8862) (5 mg) | Finerenone (BAY94-8862) (7.5 mg) | Finerenone (BAY94-8862) (10 mg) | Finerenone (BAY94-8862) (15 mg) | Finerenone (BAY94-8862) (20 mg) | Placebo
Number analyzed (Participants) | 89 | 84 | 87 | 89 | 88 | 113 | 109 | 89
scores on a scale | -2.116 (-4.521) [-4.521 to 0.289] | 0.104 (-2.369) [-2.369 to 2.577] | -1.229 (-3.643) [-3.643 to 1.185] | -1.185 (-3.597) [-3.597 to 1.226] | -2.596 (-5.049) [-5.049 to -0.142] | 0.112 (-2.054) [-2.054 to 2.278] | 0.058 (-2.146) [-2.146 to 2.263] | 0.747 (-1.684) [-1.684 to 3.178]
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) (1.25 mg) vs Placebo; Test type: Other; p = 0.0757, t-test, 2 sided; Least square mean difference = -2.863, 95% CI 2-sided [-6.022 to 0.297]
Statistical Analysis 2: Comparison: Finerenone (BAY94-8862) (2.5 mg) vs Placebo; Test type: Other; p = 0.6941, t-test, 2 sided; Least square mean difference = -0.643, 95% CI 2-sided [-3.851 to 2.565]
Statistical Analysis 3: Comparison: Finerenone (BAY94-8862) (5 mg) vs Placebo; Test type: Other; p = 0.2228, t-test, 2 sided; Least square mean difference = -1.976, 95% CI 2-sided [-5.155 to 1.203]
Statistical Analysis 4: Comparison: Finerenone (BAY94-8862) (7.5 mg) vs Placebo; Test type: Other; p = 0.2313, t-test, 2 sided; Least square mean difference = -1.932, 95% CI 2-sided [-5.098 to 1.234]
Statistical Analysis 5: Comparison: Finerenone (BAY94-8862) (10 mg) vs Placebo; Test type: Other; p = 0.0386, t-test, 2 sided; Least square mean difference = -3.342, 95% CI 2-sided [-6.509 to -0.176]
Statistical Analysis 6: Comparison: Finerenone (BAY94-8862) (15 mg) vs Placebo; Test type: Other; p = 0.677, t-test, 2 sided; Least square mean difference = -0.634, 95% CI 2-sided [-3.624 to 2.355]
Statistical Analysis 7: Comparison: Finerenone (BAY94-8862) (20 mg) vs Placebo; Test type: Other; p = 0.6536, t-test, 2 sided; Least square mean difference = -0.688, 95% CI 2-sided [-3.699 to 2.322]

5. Secondary Outcome: Change From Baseline to Day 90 in EQ-5D Scores (EQ5D - Visual Analog Scale)
Description: EuroQol Group 5-Dimension, 3-Level (EQ-5D-3L) questionnaires consist of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS was analyzed for this endpoint and it ranges from 0 (worst possible health state) to 100 (best possible health state).
Time Frame: Baseline and Day 90±2
Population: Participants in FAS with valid data for this endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862) (2.5 mg) | Finerenone (BAY94-8862) (5 mg) | Finerenone (BAY94-8862) (7.5 mg) | Finerenone (BAY94-8862) (10 mg) | Finerenone (BAY94-8862) (15 mg) | Finerenone (BAY94-8862) (20 mg) | Placebo
Number analyzed (Participants) | 89 | 83 | 86 | 89 | 86 | 112 | 109 | 88
scores on a scale | 1.381 (-1.22) [-1.22 to 3.982] | 3.888 (1.208) [1.208 to 6.568] | 3.124 (0.494) [0.494 to 5.754] | 2.851 (0.241) [0.241 to 5.461] | 2.698 (0.026) [0.026 to 5.37] | 2.743 (0.394) [0.394 to 5.092] | 1.914 (-0.465) [-0.465 to 4.292] | 4.425 (1.794) [1.794 to 7.057]
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) (1.25 mg) vs Placebo; Test type: Other; p = 0.0816, t-test, 2 sided; Least square mean difference = -3.044, 95% CI 2-sided [-6.471 to 0.383]
Statistical Analysis 2: Comparison: Finerenone (BAY94-8862) (2.5 mg) vs Placebo; Test type: Other; p = 0.7625, t-test, 2 sided; Least square mean difference = -0.537, 95% CI 2-sided [-4.027 to 2.953]
Statistical Analysis 3: Comparison: Finerenone (BAY94-8862) (5 mg) vs Placebo; Test type: Other; p = 0.4603, t-test, 2 sided; Least square mean difference = -1.301, 95% CI 2-sided [-4.759 to 2.157]
Statistical Analysis 4: Comparison: Finerenone (BAY94-8862) (7.5 mg) vs Placebo; Test type: Other; p = 0.3678, t-test, 2 sided; Least square mean difference = -1.574, 95% CI 2-sided [-5.004 to 1.855]
Statistical Analysis 5: Comparison: Finerenone (BAY94-8862) (10 mg) vs Placebo; Test type: Other; p = 0.3279, t-test, 2 sided; Least square mean difference = -1.727, 95% CI 2-sided [-5.191 to 1.736]
Statistical Analysis 6: Comparison: Finerenone (BAY94-8862) (15 mg) vs Placebo; Test type: Other; p = 0.3102, t-test, 2 sided; Least square mean difference = -1.682, 95% CI 2-sided [-4.935 to 1.57]
Statistical Analysis 7: Comparison: Finerenone (BAY94-8862) (20 mg) vs Placebo; Test type: Other; p = 0.1317, t-test, 2 sided; Least square mean difference = -2.511, 95% CI 2-sided [-5.778 to 0.755]

ADVERSE EVENTS:
Time Frame: Up to approximately 93 days after the start of study drug
Groups:
- Finerenone (BAY94-8862)(2.5 mg): 2.5 mg BAY94-8862 tablet once daily in the morning for 90 days
- Finerenone (BAY94-8862)(5 mg): 5 mg BAY94-8862 tablet once daily in the morning for 90 days
- Finerenone (BAY94-8862)(7.5 mg): 7.5 mg BAY94-8862 tablet once daily in the morning for 90 days
- Finerenone (BAY94-8862)(10 mg): 10 mg BAY94-8862 tablet once daily in the morning for 90 days
- Finerenone (BAY94-8862)(15 mg): 15 mg BAY94-8862 tablet once daily in the morning for 90 days
- Finerenone (BAY94-8862)(20 mg): 20 mg BAY94-8862 tablet once daily in the morning for 90 days
Arm/Group | Finerenone (BAY94-8862) (1.25 mg) | Finerenone (BAY94-8862)(2.5 mg) | Finerenone (BAY94-8862)(5 mg) | Finerenone (BAY94-8862)(7.5 mg) | Finerenone (BAY94-8862)(10 mg) | Finerenone (BAY94-8862)(15 mg) | Finerenone (BAY94-8862)(20 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/92 | 0/100 | 0/97 | 0/98 | 1/125 | 0/119 | 1/94
Serious Adverse Events (participants affected / at risk) | 5/96 | 3/92 | 7/100 | 8/97 | 2/98 | 6/125 | 4/119 | 3/94
Other Adverse Events (participants affected / at risk) | 14/96 | 7/92 | 13/100 | 11/97 | 10/98 | 11/125 | 12/119 | 8/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (BAY94-8862) (1.25 mg) (N=96) | Finerenone (BAY94-8862)(2.5 mg) (N=92) | Finerenone (BAY94-8862)(5 mg) (N=100) | Finerenone (BAY94-8862)(7.5 mg) (N=97) | Finerenone (BAY94-8862)(10 mg) (N=98) | Finerenone (BAY94-8862)(15 mg) (N=125) | Finerenone (BAY94-8862)(20 mg) (N=119) | Placebo (N=94)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (BAY94-8862) (1.25 mg) (N=96) | Finerenone (BAY94-8862)(2.5 mg) (N=92) | Finerenone (BAY94-8862)(5 mg) (N=100) | Finerenone (BAY94-8862)(7.5 mg) (N=97) | Finerenone (BAY94-8862)(10 mg) (N=98) | Finerenone (BAY94-8862)(15 mg) (N=125) | Finerenone (BAY94-8862)(20 mg) (N=119) | Placebo (N=94)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 3 (4) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4) | 8 (8) | 9 (9) | 5 (5) | 4 (4) | 8 (9) | 5 (6)
Dizziness (Nervous system disorders) | 6 (6) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 5 (5) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other